CLINICAL TRIAL: NCT06652100
Title: Establishment of ProNephro AKI (NGAL) Cut Off Value for Risk Assessment of Moderate to Severe Acute Kidney Injury in Adults (EPACRA-AKI)
Brief Title: Establishment of ProNephro AKI (NGAL) Cut Off Value for Risk Assessment of Moderate to Severe Acute Kidney Injury in Adults
Acronym: EPACRA-AKI
Status: Active, not recruiting | Type: Observational
Sponsor: BioPorto Diagnostics (Industry)
Collaborators: ProPharma Group (Industry)
Responsible Party: Sponsor
Other Study IDs: TD-0475
Record Dates: First submitted 2024-10-04; First posted 2024-10-22 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-11

CONDITIONS: Acute Kidney Injury
Keywords: NGAL; ICU; adult
MeSH Terms: conditions — Acute Kidney Injury

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — urine and plasma
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

INTERVENTIONS:
Diagnostic Test: ProNephro AKI (NGAL) — ProNephro AKI™ (NGAL) is an immunoassay for the in vitro quantitative determination of neutrophil gelatinase-associated lipocalin (NGAL) in human urine.

SUMMARY:
The purpose of this research is to collect blood and urine from adult patients admitted to an intensive care unit. This is to assess the performance of the ProNephro AKI (NGAL) assay (lab test) as an aid to identify patients at risk for acute kidney injury.

ELIGIBILITY:
Inclusion Criteria:

Male and females ≥ 22 years of age. Subjects must be admitted to an Intensive Care Unit and must have a urine sample collected within 24 hours of ICU admission.

Subjects must have at least one of the following leading to admission to the ICU, or occurring within 24 hours of admission to the ICU:

* Vasoactive medication administration
* Mechanical ventilation
* Hypoxemia requiring oxygen support therapy including Bilevel positive airway pressure (BIPAP) and high flow nasal canula
* Mean arterial pressure (MAP) less than 60 (within 12 hrs. of ICU admission only)
* Serum Lactate greater than 2.5 mmol/L
* History of solid organ transplantation, renal transplantation included only if more than 3 months prior
* History of bone marrow transplantation Subject with signed informed consent.

Exclusion Criteria:

Special populations including pregnant and lactating women, prisoners, or institutionalized individuals.

Subjects receiving Kidney Replacement Therapy in the first 24 hours of ICU admission.

Subjects diagnosed with active Urinary Tract Infection per institute standard of care at the time of NGAL sampling.

Subjects with a known history of chronic kidney disease stages 4 and 5 as evidenced by a pre-enrollment estimated GFR of less than 30 mL/min/1.73M2 and under the care of a nephrologist.

Subjects with any known urothelial, urological or kidney malignancies. Subjects that have had any urologic procedure or urologic surgery immediately prior to admission to the ICU.

Subjects that have had surgical nephrectomy less than 3 months prior to admission.

Subjects that have been previously enrolled in this study. Subjects that do not have a baseline sCR within 6 months prior to ICU admission available.

Subjects that did not sign the informed consent. Subjects enrolled in an interventional pharmaceutical or device clinical trial at time of ICU admission

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients admitted to the ICU 22 years of age and older
Sampling Method: Non-Probability Sample
Enrollment: 800 (Estimated)
Dates: Start 2024-10-28 (Actual); Primary Completion 2026-01-30 (Estimated); Study Completion 2026-01-31 (Estimated)

PRIMARY OUTCOMES:
Cut off Establishment | 24hrs after ICU admission
  The primary objective is to establish the cut-off value for the ProNephro AKI (NGAL) in critically ill adult patients (age 22 and older) admitted to ICU when used as an aid in risk assessment of the development of moderate to severe acute kidney injury (KDIGO stage 2/3) within 48-72 hrs. after admission.

SECONDARY OUTCOMES:
Sub-Group analysis | 24hrs after ICU admission
  Secondary objective is to explore independent cut-offs and estimate performance for NGAL in urine for the following patient subgroups:
  Patients after cardiac surgery Patients with decompensating cirrhosis Patients with sepsis Male vs female subjects Sensitivity, specificity, negative and positive predictive values are to be calculated as applicable.

CONTACTS AND LOCATIONS:
Locations (12):
- United States (12):
  - The University of Alabama, Birmingham, Alabama
  - UC Davis, Sacramento, California
  - Yale University, New Haven, Connecticut
  - University of Chicago, Chicago, Illinois
  - Johns Hopkins University, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - University of New Mexico, Albuquerque, New Mexico
  - Columbia University, New York, New York
  - Wake Forest University, Winston-Salem, North Carolina
  - Cleveland Clinic, Cleveland, Ohio
  - Medical University of South Carolina, Charleston, South Carolina

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Strader M, Imran S, Tariq A, Fraser C, Saghie E, Louis BC, Meade T, Stoyanov V, Cote JM, Twomey PJ, Murray PT. Clinical Implementation of Urinary Neutrophil Gelatinase-Associated Lipocalin Testing for Diagnosing Acute Kidney Injury in an Academic Tertiary Care Medical Centre. Kidney360. 2025 Dec 1;6(12):2119-2129. doi: 10.34067/KID.0000000887. Epub 2025 Aug 13. PMID 40802457